CLINICAL TRIAL: NCT00717210
Title: NOA-04 Randomized Phase III Study of Sequential Radiochemotherapy of Anaplastic Glioma With PCV or Temozolomide
Brief Title: Randomized Phase III Study of Sequential Radiochemotherapy of Anaplastic Glioma With PCV or Temozolomide
Acronym: NOA-04
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neuro-Oncology Working Group of the German Cancer Society (Network)
Collaborators: University Hospital Tuebingen (Other); Heinrich-Heine University, Duesseldorf (Other); Heidelberg University (Other); Charite University, Berlin, Germany (Other); University Hospital, Essen (Other); University of Leipzig (Other); University Hospital, Bonn (Other); German Cancer Research Center (Other); University of Zurich (Other)
Responsible Party: Prof. Dr. Michael Weller, NOA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOA-04
Record Dates: First submitted 2008-07-15; First posted 2008-07-17 (Estimated); Last update posted 2008-07-17 (Estimated); Status verified 2008-07

CONDITIONS: Anaplastic Astrocytoma; Oligodendroglioma; Oligoastrocytoma
Keywords: 1p/19q loss; MGMT; prognostic factors; PCV; temozolomide
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Conventional Radiotherapy
  Interventions: Radiation: Focal radiotherapy
- B1/2 (Experimental): 1:1 randomization between temozolomide and procarbazine/lomustine/vincristine (PCV)
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — 200 mg/m2 body surface on days 1-5 every 28 days for 8 cycles; and again for another 4 cycles at primary progression
  Arms: B1/2
Radiation: Focal radiotherapy — 54-60 Gy in 28-30 fractions over 6-7 weeks
  Arms: A

SUMMARY:
Background: The optimal treatment of anaplastic gliomas is controversial. Standard of care in most centers is still radiotherapy. This phase III study compared the efficacy and safety of radiotherapy vs chemotherapy in patients (pts) with newly-diagnosed, supratentorial gliomas of WHO grade III.

Methods: Pts were randomized 2:1:1 between June 1999 and February 2005 in 34 German centers to receive (i) a 6-week course of radiotherapy (1,8-2 Gy fractions, total dose 54-60 Gy) or (ii) four 6-week cycles of CCNU at 110 mg mg/m2 on day 1, vincristine at 2 mg on days 8 and 29 and procarbazine at 60 mg/m2 on days 8-21 or eight 4-week cycles of 200 mg/m2 temozolomide on days 1-5. Treatment was stopped prematurely at disease progression or occurrence of unacceptable toxicity. At this time or at disease progression, treatment in the radiotherapy group was continued with one of the chemotherapies (1:1 randomization) and with radiotherapy in both chemotherapy groups. The primary endpoint was time-to-treatment-failure (TTF) defined as progression after radiotherapy and one chemotherapy in either sequence, or any time before if further therapy could not be employed. Assuming a 50% improvement in TTF of starting with chemotherapy, 318 pts were to be enrolled to provide 80% power to achieve statistical significance at a one-sided level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* centrally confirmed anaplastic glioma according to the WHO-classification 1998/2000
* age ≥ 18 years
* Karnofsky performance status (KPS) of 70 or higher
* no prior systemic chemotherapy or radiation therapy of the brain
* no HIV infection
* adequate bone marrow reserve, liver function, and renal function
* Patients on corticosteroids had to be on a stable or decreasing dosage within the 14 days prior to randomization

Exclusion Criteria:

* Glioblastoma
* infratentorial localization of the tumor
* pregnancy or lactation period
* serious medical or neurological comorbidity
* additional malignancy requiring radio- or chemotherapy
* known hypersensitivity against study drugs
* inability to swallow
* frequent emesis
* psychological. familial, sociological or geographical situations impairing compliance with F/U examinations
* parallel participation in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 1999-06; Primary Completion 2005-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Time-to-treatment-failure defined as progression after radiotherapy and one chemotherapy in either sequence | 1999-2008

SECONDARY OUTCOMES:
Progression-free survival Overall Survival Toxicity Response rates | 1999-2012

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weller, MD, Principal Investigator — Department of Neurology, University of Zurich, Switzerland; Wolfgang Wick, MD, Study Director — Department of Neurooncology, University of Heidelberg
Locations (12):
- Germany (12):
  - University of Heidelberg, Heidelberg, Baden-Wurttemberg
  - Neurology and Radiotherapy, Tübingen, Baden-Wurttemberg
  - Klinikum Aschaffenburg, Aschaffenburg
  - Nervenklinik, Bamberg
  - Charite, Berlin
  - Neurosurgery, Düsseldorf
  - Radiotherapy, Erlangen
  - Neurology, Essen
  - Neurosurgery, Frankfurt
  - Neurosurgery, Kiel
  - Neurosurgery, Mainz
  - County District Hospital, Regensburg

REFERENCES:
- [Result] Wick W, Weller M for the Neurooncology Working Group (NOA) of the German Cancer Society Randomized phase -III study of sequential radiochemotherapy of oligoastrocytic tumors of WHO-grade III with PCV or temozolomide: NOA-04. J Clin Oncol 2008;26(15S):2007.
- [Derived] Wick W, Roth P, Hartmann C, Hau P, Nakamura M, Stockhammer F, Sabel MC, Wick A, Koeppen S, Ketter R, Vajkoczy P, Eyupoglu I, Kalff R, Pietsch T, Happold C, Galldiks N, Schmidt-Graf F, Bamberg M, Reifenberger G, Platten M, von Deimling A, Meisner C, Wiestler B, Weller M; Neurooncology Working Group (NOA) of the German Cancer Society. Long-term analysis of the NOA-04 randomized phase III trial of sequential radiochemotherapy of anaplastic glioma with PCV or temozolomide. Neuro Oncol. 2016 Nov;18(11):1529-1537. doi: 10.1093/neuonc/now133. Epub 2016 Jul 1. PMID 27370396